CLINICAL TRIAL: NCT04404530
Title: Palynziq and PKU: Treatment Impacts on Diet Quality, Neurological Health, Nutritional Status, and the Metabolome
Brief Title: Nutritional Impacts of Palynziq on Patients With Phenylketonuria (PKU)
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Rani Singh, Professor, Emory University
Other Study IDs: IRB00111450; 2025P011579 (Other: Emory IRB)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained to measure amino acids, vitamins, fats, and neurotransmitters. Blood spots will be obtained to determine the PAH gene mutation of participants.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Palynziq Therapy for PKU: Participants with PKU who are starting Palynziq therapy, or have recently started Palynziq therapy but have not achieved response.
  Interventions: Drug: Palynziq

INTERVENTIONS:
Drug: Palynziq — Participants will take Palynziq as prescribed by their genetics doctor. In accordance with the Palynziq Risk Evaluation and Mitigation Strategy (REMS) protocol, patients will have their first injection of Palynziq at the Emory Genetics Clinic under the supervision of a physician. After initiating therapy, patients will continue to mail in blood spot filter papers and 3-day dietary records to their clinic providers as standard components of clinical care.
  Other Names: Pegvaliase

SUMMARY:
Phenylketonuria (PKU) is an inherited metabolic disorder that impairs the metabolism of the essential amino acid phenylalanine (Phe). Without stringent dietary control, Phe accumulates in the blood and brain of PKU patients, leading to severe cognitive deficits. Achieving metabolic control, defined as blood Phe levels within the range of 120-360 μmol/L, has been a significant challenge for PKU patients using traditional diet therapy. The new FDA approved pharmacologic treatment, Palynziq, offers a new approach that could significantly reduce the burden of PKU by improving blood Phe levels and allowing for a less restrictive diet. As little is known about the global metabolic and physiologic effects of Palynziq, the present study aims to capture changes in diet quality, neurological health, nutritional status, the nutritional metabolome, and patient perceptions of mental and social health with sustained Palynziq therapy.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) is an autosomal recessive disorder caused by more than 500 pathogenic variants in the phenylalanine hydroxylase (PAH) gene. Due to these mutations, affected individuals have reduced activity or complete deficiency of the enzyme phenylalanine hydroxylase, which metabolizes the essential amino acid phenylalanine (Phe) to tyrosine. Consequently, Phe and its byproducts accumulate in the blood and brain of PKU patients, which can have irreparable physical and neurocognitive effects. These may include intellectual disabilities, seizures, eczema, psychosis, and hypopigmentation. To prevent these adverse conditions, early diagnosis and meticulous control of blood Phe levels are required. For optimal metabolic control, the American College of Medical Genetics (ACMG) recommends lifelong maintenance of Phe concentrations within the range of 120-360 μmol/L.

Diet therapy has dramatically improved metabolic control and nutritional status in PKU patients and when adherent to dietary treatment, numerous patients have been able to achieve normal growth and prevent severe cognitive deficits. This, however, is not an easy task given a steep restriction of intact protein is required to keep blood Phe levels within the therapeutic range. To meet nutritional needs in the absence of dietary protein, patients consume large volumes of Phe-free amino acid formulas (medical food) and specialized low-protein modified foods. While this regimen may improve overall diet quality, due to the fortification of formula with vitamins and minerals, the poor palatability and high cost medical food makes diet therapy a significant burden for patients and their families.

Pharmacologic therapies now provide an innovative approach to improve patient health and quality of life by liberalizing the traditional protein-restricted diet. Palynziq is a PEGylated recombinant of phenylalanine lyase, which can lower blood Phe concentrations. Given increasing numbers of PKU patients will be initiating Palynziq therapy, it is essential to prospectively evaluate the impact of this novel treatment on the neurological health, diet quality, and nutritional metabolome of patients when administered in a clinical setting. This knowledge will not only improve the efficacy of the treatment, but will be essential for expanding the current dietary guidelines to meet the unique needs of patients treated with Palynziq.

The objectives of this proposal are to obtain information on the diet quality, neurological health, and nutritional metabolome of patients with PKU at baseline and after intervention with Palynziq. This is a three-year observational study that includes non-pregnant adults who have PKU and have obtained a physician's prescription to initiate Palynziq treatment. Patients who complete the three year study are now eligible to participate in a sub-study which extends the main protocol for up to five years.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older
* diagnosed with PKU through newborn screening or via diagnosis later in life
* capable of providing consent for medical tests and procedures
* prescription for Palynziq and be enrolled in the Palynziq Risk Evaluation and Mitigation Strategy (REMS) program
* Substudy: Participants must have completed visit 2 of the main study

Exclusion Criteria:

* unable to provide consent
* a diagnosis of, or take medication for psychiatric, behavioral, or other inherited metabolic disorders

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with PKU
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Intra-subject Change in Intact Protein Intake | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Intra-subject change in intact protein intake will be assessed by participant-reported 3-day dietary records.
Intra-subject Change in Medical Food Protein Intake | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Intra-subject change in medical food protein intake will be assessed by participant-reported 3-day dietary records.
Sub study: Intra-subject change in intact protein and medical food protein intake. | 12 Months Post-Response through additional five years (6 years post-response)
  Intra-subject change in medical food protein intake will be assessed by participant-reported 3-day dietary records.

SECONDARY OUTCOMES:
Change in Average Intact Protein Intake | Baseline, Response (up to 60 days) 12 Months Post-Response (up to 14 months after baseline)
  Average intact protein intake will be determined by participant-reported 3-day dietary records.
Days From Palynziq Initiation to Response | Baseline up to Response (up to 60 days)
  The average length of time (in days) from Palynziq initiation until response, as defined by three consecutive plasma Phe levels lower than the upper limit of the recommended treatment range (<360 μmol/L) and a significant increase in intact protein intake (at least 60 percent of the dietary reference intake (DRI) or a two-fold increase from baseline diet prescription), will be determined.
Days From Palynziq Initiation to Consumption of Dietary Reference Intake for Intact Protein | Baseline up to 12 Months Post-Response (up to 14 months after baseline)
  The average length of time (in days) from Palynziq initiation it takes for participants to consume the dietary reference intake for intact protein (46g females, 56g males).
Change in Neuro-QOL - Cognitive Function - Short Form Score | Baseline, Response (up to 60 days) 12 Months Post-Response (up to 14 months after baseline)
  The Neuro-QOL Cognitive Function Short Form includes 8 items asking participants about their cognition during the past 7 days. Responses to statements of if cognition problems are occurring are given on a scale from 1 to 5 where 1 = very often and 5 = never. The amount of difficulty experienced from daily life tasks are responded to on a scale from 1 to 5 as 1 = cannot do task and 5 = no difficulty. Scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent in experiencing more cognition problems than the average person.
Change in Neuro-QOL Sleep Disturbance - Short Form Score | Baseline, Response (up to 60 days) 12 Months Post-Response (up to 14 months after baseline)
  The Neuro-QOL Sleep Disturbance Short Form includes 8 items asking participants about their sleep during the past 7 days. Responses to statements of if sleep problems are occurring are given on a scale from 1 to 5 where 1 = never and 5 = always. Scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent in experiencing more sleep problems than the average person.
Change in The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Score | Baseline, Response (up to 60 days) 12 Months Post-Response (up to 14 months after baseline)
  The PROMIS Global Health instrument includes 10 items asking participants about their health and quality of life. Responses to items are given on a scale from 1 to 5 where 1 = poor and 5 = excellent. Scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent in experiencing greater quality of life than the average person.
Change in PROMIS-29 Anxiety and Depression Score | Baseline, Response (up to 60 days) 12 Months Post-Response (up to 14 months after baseline)
  The PROMIS-29 instrument includes 8 items asking participants about anxiety and depression. Responses to are given on a scale from 1 to 5 where 1 = never and 5 = always. The total summed score from these items ranges from 8 to 40 and higher scores indicate greater anxiety and depression.
Change in PROMIS Emotional Support Score | Baseline, Response (up to 60 days) 12 Months Post-Response (up to 14 months after baseline)
  The PROMIS Emotional Support instrument includes 16 items asking participants about forms of emotional support they have available. Responses to items are given on a scale from 1 to 5 where 1 = never and 5 = always. Raw scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent has greater emotional support than the average person.
Change in Plasma Neurotransmitters | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Intra-subject change in neurotransmitter analysis will be assessed using fasting blood samples.
Change in Plasma Amino Acids | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Intra-subject change in plasma amino acids will be assessed using fasting blood samples.
Change in Essential Fatty Acids | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Intra-subject change in essential acids will be assessed using fasting blood samples.
Intra-subject Change in Bone Mineral Density | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Bone mineral density will be assessed with dual-energy x-ray absorptiometry (DEXA)
Intra-subject Change in Percent Fat Body Mass | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Percent fat body mass will be assessed with DEXA.
Intra-subject Change in Percent Lean Body Mass | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Percent lean body mass will be assessed with DEXA.
Intra-subject Change in Resting Energy Expenditure | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Resting energy expenditure (kilocalories/day) from Palynziq initiation through 12 months post-response will be assessed using indirect calorimetry and self-reported activity level.
Intra-subject Change in Grip Strength | Baseline through 12 Months Post-Response (up to 14 months after baseline)
  Muscle strength will be assessed using a dynamometer, which will measure grip strength on each hand.
Sub-Study: Change in Plasma Neurotransmitters | 12 Months Post-Response through additional five years (6 years post-response)
  Intra-subject change in neurotransmitter analysis will be assessed using fasting blood samples.
Sub-Study: Change in Neuro-QOL - Cognitive Function - Short Form Score | 12 Months Post-Response through additional five years (6 years post-response)
  The Neuro-QOL Cognitive Function Short Form includes 8 items asking participants about their cognition during the past 7 days. Responses to statements of if cognition problems are occurring are given on a scale from 1 to 5 where 1 = very often and 5 = never. The amount of difficulty experienced from daily life tasks are responded to on a scale from 1 to 5 as 1 = cannot do task and 5 = no difficulty. Scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent in experiencing more cognition problems than the average person.
Sub-Study: Change in Neuro-QOL Sleep Disturbance - Short Form Score | 12 Months Post-Response through additional five years (6 years post-response)
  The Neuro-QOL Sleep Disturbance Short Form includes 8 items asking participants about their sleep during the past 7 days. Responses to statements of if sleep problems are occurring are given on a scale from 1 to 5 where 1 = never and 5 = always. Scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent in experiencing more sleep problems than the average person.
Sub-Study: Change in The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Score | 12 Months Post-Response through additional five years (6 years post-response)
  The PROMIS Global Health instrument includes 10 items asking participants about their health and quality of life. Responses to items are given on a scale from 1 to 5 where 1 = poor and 5 = excellent. Scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent in experiencing greater quality of life than the average person.
Sub-Study: Change in PROMIS-29 Anxiety and Depression Score | 12 Months Post-Response through additional five years (6 years post-response)
  The PROMIS-29 instrument includes 8 items asking participants about anxiety and depression. Responses to are given on a scale from 1 to 5 where 1 = never and 5 = always. The total summed score from these items ranges from 8 to 40 and higher scores indicate greater anxiety and depression.
Sub-Study: Change in PROMIS Emotional Support Score | 12 Months Post-Response through additional five years (6 years post-response)
  The PROMIS Emotional Support instrument includes 16 items asking participants about forms of emotional support they have available. Responses to items are given on a scale from 1 to 5 where 1 = never and 5 = always. Raw scores are scaled to a T-score with a mean of 50 and a standard deviation of 10. Scores higher than 50 indicate that the respondent has greater emotional support than the average person.

CONTACTS AND LOCATIONS:
Overall Officials: Rani Singh, PhD, RDN, LD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Georgia Clinical Research Center, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No